CLINICAL TRIAL: NCT03620955
Title: Risk-stratified Therapy Based on Molecular and Cytogenetic Aberration and Treatment Response in Acute Myeloid Leukemia
Brief Title: Risk-stratified Therapy Based on Molecular Cytogenetic Aberration and Treatment Response in AML
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Second Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangzhou First People's Hospital (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Shenzhen Hospital of Southern Medical University (Other); Peking University Shenzhen Hospital (Other); Shenzhen Second People's Hospital (Other); Zhongshan People's Hospital, Guangdong, China (Other); First Affiliated Hospital of Guangxi Medical University (Other); Xiangya Hospital of Central South University (Other); The Third Xiangya Hospital of Central South University (Other); First Affiliated Hospital of Gannan Medical University (Other); Peking University People's Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Affiliated Hospital of Zhengzhou University (Other); Chenzhou NO. 1 people's Hospital (Unknown)
Responsible Party: Principal Investigator, Qifa Liu, professor, Nanfang Hospital, Southern Medical University
Other Study IDs: Risk stratification in AML
Record Dates: First submitted 2018-08-05; First posted 2018-08-08 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Risk-directed Therapy; Cytogenetic Abnormality; Molecular Abnormality; MRD
MeSH Terms: conditions — Chromosome Aberrations; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Risk stratification: Risk stratification based on cytogenetic and molecular and MRD level after three courses of chemo therapy.
  Interventions: Other: Justified risk stratification based on MRD after three course chemo therapy

INTERVENTIONS:
Other: Justified risk stratification based on MRD after three course chemo therapy — All patients are routinely divided into different risk groups according to the NCCN guild based on cytogenetic and molecular abnormality. Then all patients are treated with anthracycline combined with cytarabine regimens for two courses . The patients without obtaining CR will go on one cycle of salvage therapy and then be bridged to allo-HSCT. Those acquiring CR will be given one more course of HDAC as consolidation treatment and then be detested MRD with flow cytometry after that. The patients with MRD positive would be moved to a higher risk class.The stratified therapy should be considered according to the new risk stratification.

SUMMARY:
Risk-stratified therapy based on molecular and cytogenetic for acute myeloid leukemia (AML) is well accepted and benefits patients' survival. However, neither every patient with low risk factors obtains better survival, nor all high risk patients experience worse outcome. Lots of data have shown that the early treatment response presenting as minimal residual disease (MRD) has an important role in prognostic prediction. In this study, we perform risk stratification based on not only Cytogenetic and Molecular characteristic, but also MRD after three courses of chemo therapy in AML cohort. Patients with MRD positive would be moved to a higher risk class. And then the risk-stratified therapy should be considered according to the new risk stratification.

DETAILED DESCRIPTION:
Risk-stratified therapy based on cytogenetic and molecular characteristic for acute myeloid leukemia (AML) is well accepted and benefits patients' survival. However, neither every patient with low risk factors obtains better survival, nor all high risk patients experience worse outcome. Lots of data have shown the important role of early treatment response presenting as minimal residual disease (MRD) in prognostic prediction. In this study, we perform risk stratification based on not only cytogenetic and molecular characteristic, but also MRD levels after three courses of chemo therapy. We stratified all patients into different risk groups according to the NCCN guild based on cytogenetic and molecular. Then we treat all patients with anthracycline combined with cytarabine regimens for two courses (First cycle: IDA 12mg/m2 or DNR 60mg/m2, d1-3, Ara-C 100mg/m2 d1-7; Second cycle: IDA 10mg/m2 or DNR 45mg/m2, d1-3, Ara-C 2g/m2 q12h, d1-3) . The patients without obtaining complete remission (CR) will go on one cycle of salvage therapy and then be bridged to allogeneic (allo-) hemopoietic stem cell transplantation (HSCT). Those acquiring CR will be given one course of high dose cytarabine (HDAC) as consolidation treatment and then be detested MRD with flow cytometry after that. The patients with MRD positive would be moved to a higher risk class.The stratified therapy should be considered according to the new risk stratification.The patients with MRD negative in low risk group are given HDAC (Ara-C 2g/m2 q12h, d1-3) for 3 cycles. If MRD is continuously negative in this cohort, chemotherapy will be stopped and MRD will be continuously monitored to the third year after the diagnosis. The patients with MRD negative in medium risk group are suggested to receive allo-HSCT if a HLA-matched sibling donor is available, or autologous (auto-) HSCT after receiving HDAC regimen for one more cycle if no HLA-matched sibling donors are available. The patients with MRD positive in low or medium-risk group or the cases in high-risk group are going to be bridged into allo-HSCT if a donor is available including haploid donors. The aim of this study is to evaluate whether the new stratification system benefits AML patients with better OS and DFS.

ELIGIBILITY:
Inclusion Criteria:

All newly diagnosed AML exclusively of APL with age range from 14 to 60-year old

Exclusion Criteria:

Any abnormality in a vital sign (e.g., organ function failure, serious infection ) Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All newly diagnosed AML exclusively of APL with age range from 14 to 60-year old.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-08-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
relapse rate | 2 year

SECONDARY OUTCOMES:
overall survival (OS) | 2 year
disease-free survival (DFS) | 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Department of Hematology,Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang Y, Feng Z, Du J, Liu H, Yu S, Liang X, Zhao W, Zhang Q, Zhang X, Nie D, Sun Z, Du X, Xu X, Yu G, Shi P, Liu Q, Shao R, Qu H, Xiong W, Wang S, Jiang Y, Zhang H, Guo Z, Dai M, Jiang X, Xu D, Huang F, Fan Z, Xu N, Liu C, Wu M, Lin R, Jin H, Sun J, Liu Q, Xuan L. High-dose cytarabine with idarubicin consolidation for acute myeloid leukemia in first complete remission: a randomized controlled trial. Leukemia. 2025 Aug;39(8):1857-1864. doi: 10.1038/s41375-025-02655-x. Epub 2025 May 28. PMID 40437173